CLINICAL TRIAL: NCT06436924
Title: Safety and Efficacy of Workflows of High Volume Single Operators in a Left Atrial Appendage Occlusion Device Implant Procedural Day: SAFE HV
Brief Title: Safety and Efficacy of Workflows of High Volume Single Operators in a LAAO Device Implant Procedural Day
Status: Recruiting | Type: Observational
Sponsor: Heart Rhythm Clinical and Research Solutions, LLC (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: SAFE HV
Record Dates: First submitted 2024-05-22; First posted 2024-05-31 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Subjects undergoing LAAO device implant: Watchman LAAO device implant
  Interventions: Device: Left Atrial Appendage Device Implant

INTERVENTIONS:
Device: Left Atrial Appendage Device Implant — The Watchman Device is implanted into the left atrial appendage and is designed to close it off and keep blood clots from escaping that area.

SUMMARY:
SAFE HV is an observational, prospective, multi-center, non-randomized study evaluating real-world clinical experience of centers where a single procedural physician schedules eight or more left atrial appendage occlusion (LAAO) device implant procedures in a single calendar day.

DETAILED DESCRIPTION:
Since 2009, Watchman FLX™ and its predecessor, Watchman™ have provided a safe and effective alternative to oral anticoagulation for over 200,000 patients in the United States and Europe. Advancements in the design of the Watchman FLX™ have made the device available to a wider range of patients. As more patients qualify for the device, more implant procedures are necessary to provide them with this life-changing treatment option.

Some Watchman FLX™ implanters perform high volumes of implant procedures on certain days. While performing a high-volume of implant procedures is desirable for many reasons, it must be determined that cases performed under such circumstances are comparable in safety and efficacy to implant procedures performed at lower volumes. While there has been no differentiation between high and low volume cases in previous studies, data obtained in this study will be compared to overall safety and efficacy data available from the PINNACLE FLX clinical trial and the SURPASS analysis to ensure that safety and efficacy outcomes are comparable.

Additionally, this study will collect data on the workflows of these high-volume implanters that will help determine which factors contribute to the successful performance of high volumes of Watchman FLX™ implants in a single day. In the future this information may be used to help other implanters optimize workflows to increase their volume of daily implants and hence, provide more opportunities for patients to access this transformative device.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Able and willing to participate in baseline and follow up evaluations for the full length of the study
3. Clinically qualified, in the opinion of the Investigator, to receive a LAAO device
4. Receiving a Watchman FLX™ or Watchman FLX Pro™ LAAO device as part of their plan of care
5. Having their LAAO device implant procedure scheduled on a qualifying high-volume* procedure day as assessed within 2 days (≤ 2 calendar days) prior to the planned procedure date

   *high-volume - a calendar day in which the single implanting physician schedules ≥ 8 LAAO device implant procedures, regardless of the device manufacturer
6. Willing and able to provide informed consent

Exclusion Criteria:

1. Enrolled in an investigational drug or device clinical trial, or any trial that dictates the treatment plan
2. In the opinion of the Investigator, any known contraindication to a LAAO device or implant procedure
3. Having their LAAO device implant procedure scheduled on a day in which the single implanting physician scheduled < 8 LAAO device implant procedures as assessed within 2 days (≤ 2 calendar days) prior to the planned procedure date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include subjects who are clinically qualified for a Watchman FLX™ or Watchman FLX Pro™ LAAO device implant and would receive one regardless of participation in the study, who meet all eligibility criteria for the study, and present at participating institutions for a LAAO device implant procedure on a day in which a single implanting physician scheduled at least eight LAAO device implant procedures, regardless of the device manufacturer (i.e., high-volume).
Sampling Method: Probability Sample
Enrollment: 678 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Peri-procedural complications | Procedure through discharge, an average of 1-3 days
  Incidence of peri-procedural complications summarized descriptively and compared to historical data
Peri-device leakage | Date of implant up to 90 days
  Assessed by successful closure of the left atrial appendage defined by peri-device leakage of <5mm. This will be identified at the post implant imaging.
Late onset complications | Discharge to 30 days.
  Incidence of post procedure complications summarized descriptively and compared to historical data.

CONTACTS AND LOCATIONS:
Overall Officials: Saumil Oza, MD, Principal Investigator — St. Vincent's
Locations (7):
- United States (7):
  - Grandview Medical Center, Birmingham, Alabama
  - Pima Heart and Vascular, Tucson, Arizona
  - The Medical Center of Aurora, Aurora, Colorado
  - Ascension St. Vincent, Jacksonville, Florida
  - Naples Community Hospital, Naples, Florida
  - Memorial Health University Medical Center, Savannah, Georgia
  - Medical University of South Carolina, Columbia, South Carolina